CLINICAL TRIAL: NCT04861467
Title: A Randomized, Open Study of Camrelizumab vs Placebo as a Maintenance Therapy After Chemoradiation in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Camrelizumab as a Maintenance Therapy After Chemoradiation in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jun-Lin Yi, MD, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CATCH
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: HNSCC
Keywords: Immunotherapy; Chemoradiation
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: Camrelizumab (Experimental): camrelizumab as maintenance therapy after Chemoradiation(evaluation results：PR/SD)
  Interventions: Drug: Camrelizumab
- observation (No Intervention): observation after Chemoradiation
- Exploration：Camrelizumab (Experimental): camrelizumab for maintenance after chemoradiation( evaluation results：CR)
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — IV
  Arms: Experimental: Camrelizumab; Exploration：Camrelizumab

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of Camrelizumab as maintenance therapy in newly diagnosed locally advanced head and neck squamous cell carcinoma subjects after chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

* Who have histologic or cytologic confirmation of head and neck squamous cell carcinoma in the mouth, oropharynx (p16-), hypopharynx, or larynx.
* Local advanced head and neck squamous cell carcinoma diagnosed as stage III-IVa by AJCC 8
* Except for the prescribed radical radiotherapy and chemotherapy regimen, there has been no previous treatment for LA-HNSCC systemic antitumor or local radical therapy (allowing the prescribed induction chemotherapy regimen before radical radiotherapy and chemotherapy)
* 28 days after radical radiotherapy and chemotherapy (radiotherapy and chemotherapy (±7 days) did not show disease progression, and consideration was given within 28 days after curative effect evaluation
* Clinically assessable lesions according to RECIST1.1,(lesion length ≥10 mm or lymph node short diameter ≥15 mm)
* The age at which informed consent is signed is 18-70 years, male and female
* KPS score ≥80 percent
* Estimated lifetime ≥6 months
* The function of important organs meets the following requirements (excluding the use of any blood components and cytokines within 14 days):

Normal bone marrow reserve function: WBC≥3.0×10^9/ L, NEUT≥1.5×10^9/ L, PLT≥80×10^9/ L, Hb≥90g/L Normal renal function or SCr≤1.5 times normal upper limit (ULN) or Ccr≥50 ml/min ; Normal liver function or TBIL≤1.5 times the upper limit of normal value (ULN); AST or ALT level 2.5 times the upper limit of normal value (ULN);

* Ability and willingness to follow research and follow-up procedures
* Men and women of childbearing age must agree to adequate contraception throughout the study period and within 6 months after treatment
* The subjects volunteered to join the clinical study and signed informed consent, good compliance and follow-up

Exclusion Criteria:

* 1.Have received any systemic anti-tumor therapy against the target lesion
* Previous experience in head and neck radiotherapy
* Previous immunotherapies including anti PD-1/PD-L1, anti CTLA-4, etc
* Subjects who received anti-tumor vaccines or other immunomodulatory drugs (e.g. interleukin-2, thymosin, Lentinus edodes polysaccharide, etc.) within 1 month prior to joining the group, or who received live attenuated vaccines
* Subjects who had been systematically treated with corticosteroids (prednisone or other equivalent hormones >10 mg/ days) or other immunosuppressants within 1 month of entry. To allow inhaled or local use of corticosteroids in the absence of active autoimmune disease, as well as adrenocorticotropic replacement therapy ≤10 days mg/ dose of prednisone
* Pleural effusions, pericardial effusions or ascites requiring drainage, or serosal effusions for treatment within 2 weeks prior to group entry
* No active autoimmune disease or history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitary, vasculitis, nephritis, hyperthyroidism, hypothyroidism) may be included
* Subjects with severe infection within 1 month prior to admission, including, but not limited to, infection complications requiring hospitalization, bacteremia, severe pneumonia, etc. Subjects with any active infection, or unexplained fever >38.5℃ during screening, prior to first administration
* Severe cardiovascular disease: grade II myocardial ischemia or myocardial infarction, uncontrolled arrhythmia; grade III ~ IV cardiac insufficiency, or echocardiography indicated that left ventricular ejection fraction (LVEF)<50%;
* The subjects were treated with bronchiectasis and other systemic treatments. Asthma control was unsatisfactory and could not be included (asthma was completely alleviated in childhood and included without any intervention in adults)
* HIV infection or known AIDS, active hepatitis B (HBV DNA≥500 IU/ml), hepatitis C (hepatitis C antibody positive, and HCV-RNA higher than the lower detection limit of the analytical method) or combined with hepatitis B and hepatitis C infection;
* Subjects with a history of other malignancies within five years (except complete treatment of skin cancer with cervical or basal cell carcinoma or squamous cell carcinoma in situ)
* Patients with a clear history of allergies may be allergic to, or intolerant to Camrelizumab
* Persons with a history of substance abuse and who are unable to abstain or who have mental disorders Increasing the risk associated with participating in a study or research drug and, according to the researcher's judgment, other circumstances in which the subjects are not suitable for inclusion in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
median progression-free survival(in accordance with RECIST1.1) | Up to 3 years
  mPFS is the median time from the date of randomization to the date of first record of disease progression or death.

SECONDARY OUTCOMES:
1 year progression-free survival rate | 1 year from the the date of randomization
overall survival | Up to 3 years
  OS is the time from randomization to death due to any cause.
objective response rate | Up to 3 years
disease control rate | Up to 3 years
time to progression | Up to 3 years
progression-free survival(in accordance with irRECIST1.1) | Up to 3 years

OTHER OUTCOMES:
event-free survival in exploration group | Up to 3 years
  EFS is the time from the date of randomization to any event

CONTACTS AND LOCATIONS:
Overall Officials: Junlin Yi, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer hospital, Chineses Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided